CLINICAL TRIAL: NCT00674557
Title: A Cancer Research UK Randomised Phase II Trial of ATN-224 (Copper Binding Agent) in Combination With Exemestane Versus Exemestane Alone in Post-menopausal Women With Recurrent or Advanced, Oestrogen and/or Progesterone Receptor Positive Breast Cancer
Brief Title: Exemestane With or Without ATN-224 in Treating Postmenopausal Women With Recurrent or Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn as the clinical development of ATN-224 was terminated by the drug company who was providing ATN-224 for the study
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRUK-CR0207-22; CDR0000595074 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-005752-16; EU-20850
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; HER2-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tetrathiomolybdate; exemestane

INTERVENTIONS:
Drug: SOD1 inhibitor ATN-224
Drug: exemestane
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Exemestane may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. ATN-224 may stop the growth of breast cancer by blocking blood flow to the tumor. It is not yet known whether giving exemestane together with ATN-224 is more effective than giving exemestane alone in treating patients with recurrent or advanced breast cancer.

PURPOSE: This randomized phase II trial is studying the side effects of exemestane given together with or without ATN-224 and to see how well it works in treating postmenopausal women with recurrent or advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of postmenopausal women with, estrogen receptor- and/or progesterone receptor-positive recurrent or advanced breast cancer treated with exemestane with versus without SOD1 inhibitor ATN-224.
* Establish the safety of SOD1 inhibitor ATN-224 in combination with exemestane in these patients.

Secondary

* Determine the response rate (overall, at 16 and 24 weeks), response duration, and rate of stable disease for ≥ 16 and ≥ 24 weeks in these patients.
* Determine the clinical benefit rate (complete response, partial response, and stable disease) at 16 and 24 weeks in these patients.
* Investigate the time course of suppression of serum ceruloplasmin (Cp, surrogate for copper).
* Investigate serum estradiol and estrone sulphate levels in these patients to assess if SOD1 inhibitor ATN-224 interacts with the aromatase inhibition of exemestane.

Tertiary

* Investigate the pharmacokinetic behavior of SOD1 inhibitor ATN-224 in combination with exemestane.
* Investigate superoxide dismutase 1 (SOD1) activity in red blood cells and cytokine levels in plasma samples from these patients.
* Investigate circulating endothelial cell levels, circulating endothelial RNA levels, and proteome profiles in blood samples at baseline and during treatment, from these patients.
* Investigate SOD1, lysyl oxidase and copper-dependent proteins expression, and endothelial growth factor receptor-related cell-signaling pathways in historical tumor samples from all patients entered on the study.

OUTLINE: This is a multicenter study. Patients are stratified according to prior aromatase inhibitor therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral exemestane and oral SOD1 inhibitor ATN-224 once daily.
* Arm II: Patients receive oral exemestane once daily. In both arms, treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic and pharmacodynamic assessments, including Cp levels, estradiol and estrone sulfate, SOD1 levels, cytokines, proteomics, circulating endothelial RNA, circulating endothelial cells, protein expression, and EGFR-related cell signaling pathways.

After completion of study treatment patients are followed at 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Recurrent disease after 2-3 years of adjuvant treatment with an anti-estrogen (documented by imaging techniques)
  * Advanced disease that has recurred during or after anti-estrogen therapy
* Measurable or evaluable disease by conventional techniques, with ≥ 1 lesion that can be followed for response

  * Bone metastases only are eligible provided they have ≥ 1 lytic lesion (not previously irradiated or planned for irradiation) that can be followed by X-ray or CT scanning
  * Cutaneous skin metastases only are eligible provided the skin lesions are > 10 mm and can be followed by good quality photography with a ruler included in the photograph
* No clinically apparent brain metastases
* Hormone receptor status must meet 1 of the following criteria:

  * Estrogen receptor-positivity

    * Score ≥ 3 on a scale (range of 0 to 8), or equivalent score from other grading methods, representing the intensity and percentage of positive-staining tumor cells by immunohistochemistry
    * Greater than or equal to 5 fmol/mg protein by ligand binding assay or ELISA
  * Progesterone receptor-positivity

    * Score ≥ 3 on a scale (range of 0 to 8) or equivalent score from other grading methods, representing the intensity and percentage of positive-staining tumor cells by immunohistochemistry
* No HER-2 overexpression, defined as gene amplification by fluorescence in situ hybridization [FISH] OR 3+ overexpression by IHC)

PATIENT CHARACTERISTICS:

* Postmenopausal as defined by any of the following:

  * Surgical or radiation-induced
  * No menstrual periods for 12 consecutive months with no other biological or physiological cause in women with an intact uterus
  * Age ≥ 55 years
* WHO performance status 0-2
* Life expectancy ≥ 6 months
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and/or AST ≤ 2.5 times ULN (5 times ULN if due to tumor)
* Creatinine clearance ≥ 50 mL/min
* No history of malabsorption syndromes or other gastrointestinal disorders that may affect SOD1 inhibitor ATN-224 absorption, including any of the following:

  * Bowel obstruction
  * Celiac disease
  * Sprue
  * Cystic fibrosis
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to SOD1 inhibitor ATN-224, omeprazole (or other proton pump inhibitor), or exemestane
* No non-malignant systemic disease including active uncontrolled infection
* No serologic positivity for hepatitis B, hepatitis C, or HIV
* No concurrent congestive heart failure
* No history of NYHA class III-IV cardiac disease
* No other concurrent malignancy, except adequately treated cone-biopsied carcinoma in situ of the uterine cervix, basal cell or squamous cell carcinoma of the skin

  * Cancer survivors who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 5 years, and are deemed at low risk for recurrence are eligible
* No other condition which, in the investigator's opinion, would not make the patient a good candidate for this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy (alopecia allowed)
* At least 1 year since prior bilateral oophorectomy
* Prior adjuvant or neoadjuvant treatment with tamoxifen allowed
* Prior adjuvant therapy with a non-steroidal aromatase inhibitor allowed
* More than 4 weeks since prior immunotherapy or chemotherapy (6 weeks for nitrosoureas and mitomycin-C)
* More than 4 weeks since prior major thoracic and/or abdominal surgery
* More than 3 weeks since prior endocrine therapy
* More than 4 weeks since prior and no concurrent radiotherapy (except to control pain or prevent fracture)
* No prior exemestane
* Concurrent iron-containing vitamins or supplements are allowed
* No concurrent luteinizing hormone-releasing hormone analog
* No concurrent oral bisphosphonates (IV bisphosphonates allowed)
* No concurrent chronic steroid therapy for concurrent illness or cancer (short-term steroid use for concurrent illness allowed [e.g., for acute asthma])
* No concurrent copper- or zinc-containing vitamins or supplements
* No concurrent participation in another interventional clinical study (participation in an observational study allowed)
* No other concurrent copper-binding drug (e.g., penicillamine or trientine)
* No other concurrent anticancer therapy or investigational agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2008-06; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival
Safety

SECONDARY OUTCOMES:
Response rate (complete and partial response) overall and at 16 and 24 weeks
Rate of stable disease for ≥ 16 and ≥ 24 weeks
Response duration
Clinical benefit rate (complete and partial response, stable disease) at 16 and 24 weeks
Time (in days) taken after starting SOD1 inhibitor ATN-224 to achieve target serum ceruloplasmin level (5 to 15 mg/dl)
Levels of serum estradiol and estrone sulphate at day 1 of course 1 and 2
Molybdenum levels at single time-points at the beginning of course 1 to 6 in patients taking SOD1 inhibitor ATN-224 in combination with exemestane.
SOD1 activity in red blood cells and cytokine levels in plasma samples
Circulating endothelial cell and circulating endothelial RNA levels, and proteome profiles in blood samples at baseline and during treatment
SOD1 and lysyl oxidase expression, and copper-dependent proteins and endothelial growth factor receptor-related cell-signaling pathways in historical tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Adrian L. Harris, MD, Principal Investigator — Churchill Hospital
Locations (1):
- Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Oxford, England, United Kingdom